CLINICAL TRIAL: NCT00996515
Title: A Phase 1 Protocol of 5-Azacytidine and Erlotinib in Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0710C; NCI-2011-02646 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Solid Tumor Malignancies
Keywords: Advanced Solid Tumor Malignancies; Erlotinib; Vidaza; Tarceva; 5-azacytidine
MeSH Terms: interventions — Azacitidine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 5 (Experimental): Erlotinib 150mg/day PO Day 1-28 and Vidaza 100mg/m2/day SQ Day 1-4 and 15-18
  Interventions: Drug: 5-azacytidine, erlotinib; Drug: Erlotinib PO and Vidaza IV
- Cohort 4 (Experimental): Erlotinib 200 mg/day PO Day 1-28 and Vidaza 75 mg/m2/day SQ 1-4 and 15-18
  Interventions: Drug: 5-azacytidine, erlotinib; Drug: Erlotinib PO and Vidaza IV
- Cohort 3 (Experimental): Erlotinib 150 mg/day PO Day 1-28 and Vidaza 75 mg/m2/day IV Day 1-3 and 15-17
  Interventions: Drug: 5-azacytidine, erlotinib; Drug: Erlotinib PO and Vidaza IV
- Cohort 2 (Experimental): Erlotinib 150 mg/day PO Day 1-28 and Vidaza 75 mg/m2/day IV Day 1-2 and 15-16
  Interventions: Drug: 5-azacytidine, erlotinib; Drug: Erlotinib PO and Vidaza IV
- Cohort 1 (Experimental): Erlotinib 150 mg/day PO Day 1-28 and Vidaza 75 mg/m2/day IV Day 1 and 15
  Interventions: Drug: 5-azacytidine, erlotinib; Drug: Erlotinib PO and Vidaza IV

INTERVENTIONS:
Drug: 5-azacytidine, erlotinib — Erlotinib 150 mg PO daily, days 1-8, and 15-22 5-Azacytidine 75 mg/m2/day, IV days 1 and 15
  Other Names: Erlotinib :- Tarceva™ (OSI-774); Vidaza (5-azacytidine)
Drug: Erlotinib PO and Vidaza IV — Patients enrolled to 1 of 5 cohorts, with varying drug doses and dose scheduling.

SUMMARY:
PRIMARY OBJECTIVES:

I. To document the toxicities, and reversibility of toxicities, of this regimen of 5-azacytidine (azacitidine) and erlotinib (erlotinib hydrochloride).

SECONDARY OBJECTIVES:

I. To determine any potential anti-tumor effects, as determined by the objective tumor response (complete and partial responses), clinical benefit (complete and partial responses, and clinical benefit), the time to tumor response, the time to tumor progression, and the overall survival.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study.

Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1 and 15, days 1-2 and 15-16, days 1-3 and 15-17, or days 1-4 and 15-18. Patients also receive erlotinib hydrochloride orally (PO) daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 28 days and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfill all of the following criteria to be eligible for study entry:
* Those who will be eligible will be all patients with non-hematologic neoplasms (lymphomas, leukemias, myeloma, myelodysplasia, or myeloproliferative syndromes) who have disease which has been previously treated and/or for which there is no acceptable standard treatment regimen available, and cannot be treated definitively with either surgery or radiotherapy. All will be appropriate candidates for treatment, and are not candidates for treatment with protocols of higher priority. All patients should have an ECOG/Zubrod/SWOG performance status of <2 at the time of the initiation of therapy, adequate end-organ function, no severe comorbid disease, and ability to provide informed consent.

Other Eligibility Criteria:

* Signed Informed Consent
* ECOG/Zubrod/SWOG Performance Status <2 (Karnofsky Performance Status > 70%)
* Life expectancy > 8 weeks
* Male or female' age >18 years
* Patients of childbearing potential must be using an effective means of contraception.
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment.
* Histologic diagnosis of a solid tumor malignancy that is advanced and cannot be treated adequately by radiotherapy or surgery; or metastatic disease
* Baseline laboratory values (bone marrow, renal, hepatic):

  * Adequate bone marrow function:
  * Absolute neutrophil count >1000/µL
  * Platelet count >100'000/µL
  * Renal function:
* Serum creatinine < 1.5 x ULN

  * Hepatic function:
* Bilirubin <1.5x normal

  * Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels <=2 x ULN
  * Serum calcium < 12 mg/dl

Exclusion Criteria:

Patients meeting any of the following criteria are ineligible for study entry:

* Pregnant or lactating females
* Myocardial infarction or ischemia within the 6 months before Cycle 0' Day 0
* Uncontrolled' clinically significant dysrhythmia
* Prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* Uncontrolled metastatic disease of the central nervous system
* Sensitivity to erlotinib, 5-azacytidine or mannitol
* Advanced hepatic tumors
* Radiotherapy within the 2 weeks before Cycle 1' Day 1
* Surgery within the 2 weeks before Cycle 1' Day 1
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Quality and quantity of adverse events due to administration of erlotinib + 5-azacytidine, as therapy for the treatment of advanced or metastatic cancer. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States